CLINICAL TRIAL: NCT03183882
Title: Effect of Peer Comparison Feedback on Opioid Prescribing by Emergency Medicine Providers
Brief Title: Peer Comparison Feedback on Opioid Prescribing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Brian Suffoletto, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PRO17040547
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Opioid Use

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normative Peer Comparison (Experimental): One-time summary report of 14-month individual history of opioid prescribing WITH comparisons to (a) other providers at their site and (2) other providers at 15 ED sites with similar prescribing
  Interventions: Behavioral: Peer Normative Comparison Feedback
- Control Feedback (Active Comparator): One-time summary report of their individual history of opioid prescribing
  Interventions: Behavioral: Personal Feedback

INTERVENTIONS:
Behavioral: Personal Feedback — One-time summary report of their individual history of opioid prescribing over the past 14 months
  Arms: Control Feedback
Behavioral: Peer Normative Comparison Feedback — One-time summary report of their individual history of opioid prescribing over the past 14 months WITH comparisons to (a) other providers at their site and (2) other providers at all 15 ED sites with similar prescribing
  Arms: Normative Peer Comparison

SUMMARY:
We aim to determine if descriptive normative feedback of peer prescribing reduces opioid analgesic prescribing by emergency medicine providers

DETAILED DESCRIPTION:
State-based Prescription Drug Monitoring Programs (PDMPs) are being implemented to reduce prescription drug abuse and diversion. On August 24, 2016, Pennsylvania initiated its mandated PDMP. In prior research, we found that ED providers reduced opioid prescribing by 17% immediately after PDMP went live. Still, there is variability between providers in the frequency of opioid prescribing even after PDMP initiation. Changing clinician prescribing behavior is difficult, but recent research has shown that using peer comparisons can assist behavior change (Meeker D et al., JAMA, 2016). In this study, we will randomize a convenience sample of ED providers to receive either their opioid prescribing history data with peer comparative data or without peer comparative data. We will examine the effect on immediate perceived norms as well as impact on opioid prescribing in the subsequent 3 months. Results could inform behavioral feedback to alter clinician prescribing behaviors

ELIGIBILITY:
Inclusion Criteria:

* Emergency medicine provider
* Writes 10 or more opioid prescriptions per month (on average)

Exclusion Criteria:

* none

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2017-09-28 (Actual); Study Completion 2017-09-28 (Actual)

PRIMARY OUTCOMES:
Normative beliefs | Pre-post intervention
  How much, relative to other emergency providers, do they prescribe opioids?
Number of opioid prescriptions per month | 3-months pre-intervention to 3-months post intervention
  Number of opioid prescriptions written

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh Medical Center Emergency Department, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share